CLINICAL TRIAL: NCT00469482
Title: A Randomized Control Trial Using the BIS Monitor to Avoid Over Sedation and Prolonged Neuropsychological Deficits in Mechanically Ventilated ICU Patients
Brief Title: The SOMNUS Study: Sedative Optimization Via Monitoring Neurological Status
Acronym: SOMNUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Wes Ely, Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 061218; SOMNUS (Other: Aspect Medical Systems, Inc.)
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Delirium; Cognitive Impairment; Critically Ill
Keywords: Delirium; Cognitive Impairment; Sleep; Polysomnography; Sedation; Mechanical Ventilation; Critical Illness
MeSH Terms: conditions — Delirium; Cognitive Dysfunction; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sedation, RASS Targeted (Active Comparator): Patient sedation utilizing standard of care methods (RASS Targeted)
  Interventions: Other: Sedation, RASS Targeted
- Sedation,RASS Targeted plus BIS Monitoring (Active Comparator): Providing patient sedation utilizing standard of care methods (RASS) plus BIS monitoring.
  Interventions: Other: Sedation,RASS Targeted plus BIS Monitoring

INTERVENTIONS:
Other: Sedation,RASS Targeted plus BIS Monitoring — Providing patient sedation utilizing standard of care methods (RASS) plus BIS monitoring
  Arms: Sedation,RASS Targeted plus BIS Monitoring
Other: Sedation, RASS Targeted — Patient sedation utilizing standard of care methods (RASS targeted)
  Arms: Sedation, RASS Targeted

SUMMARY:
A combined strategy of Richmond Agitation and Sedation Scale (RASS) clinical targeting plus bispectral index (BIS) guided sedation in mechanically ventilated, critically ill patients will decrease time on mechanical ventilation, decrease the duration of intensive care unit (ICU) delirium and coma, and will improve subacute neurocognitive function when compared to sedation guided by RASS targeting alone.

DETAILED DESCRIPTION:
Sedatives and analgesics are used to maintain comfort in almost all mechanically ventilated patients. Unfortunately, these medications also have many deleterious effects. Sedatives increase time on mechanical ventilation, have adverse hemodynamic effects, disturb sleep architecture, and have been determined to be an independent risk factor for ICU delirium. Delirium is an independent determinant of longer hospital stay, higher costs, and higher mortality, and the presence of delirium is highly predictive of long-term neurocognitive deficits. In consideration of these facts, better methods are needed to guide sedation, avoid oversedation, and possibly reduce delirium.

Current guidelines recommend titration of sedation to a goal level based on bedside evaluation using a validated assessment tool, e.g. the Richmond Agitation and Sedation Scale. These assessment tools, however, are underused and many ICU patients are oversedated with well described consequences. A practical method by which to determine where a patient lies may prove beneficial in optimizing our delivery of sedatives and improving patient outcomes.

While conventional EEG monitoring is not practical in the ICU, bispectral index (BIS) monitoring may be easily used in this clinical setting. BIS monitoring may provide a means to assess sedation level in unresponsive or paralyzed ICU patients and to decrease the total amount of sedatives/analgesics administered. Additional benefits of a combined clinical sedation scale and BIS-monitoring approach could include a decreased incidence and/or duration of delirium as well as a decreased incidence and severity of ICU-associated prolonged neurocognitive deficits.

The specific aims of this study are as follows:

Aim 1: To determine if sedative and analgesic medication delivery guided by clinical sedation scales and BIS monitor parameters of over-sedation will decrease time on mechanical ventilation.

Aim 2: To determine if sedative and analgesic medication delivery guided by clinical sedation scales and BIS monitor parameters of over-sedation will decrease the duration of delirium and coma when compared to the use of clinical sedations scales alone.

Aim 3: To determine if sedative and analgesic medication delivery guided by clinical sedation scales and BIS monitor parameters of over-sedation will decrease the incidence and severity of subacute cognitive impairment when compared to the use of clinical sedation scales alone.

Aim 4: To characterize polysomnography findings in critically ill patients at various BIS levels.

Aim 5: To determine if poor sleep quality is a factor in post critical illness neurocognitive dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult patients admitted to the ICU for critical illnesses requiring mechanical ventilation with expectation of being mechanically ventilated for greater than 24 hours. Subjects must have an actual or a target RASS of -3 or deeper with 48 hours of initiation of mechanical ventilation.

Exclusion Criteria:

* Subjects who are less than 18 years old.
* Inability to obtain informed consent from the patient or his/her surrogate.
* Subjects admitted with alcohol or drug overdoses, suicide attempts, or alcohol/delirium with tremors.
* Subjects with documented moderate to severe dementia.
* Subjects with anoxic brain injuries, strokes, neurotrauma, or neuromuscular disorders such as myasthenia gravis or Guillain Barre syndrome.
* Subjects whose family and/or physician have not committed to aggressive support for 72 hours or who are likely to withdraw within 72 hours.
* Subjects who are moribund or are not expected to survive hospital discharge due to preexisting uncorrectable medical condition.
* Subjects who have either Child-Pugh Class B or C cirrhosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-06; Primary Completion 2008-10 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of ventilator free hours and days | while in ICU, appoximately 3-7 days

SECONDARY OUTCOMES:
Number of delirium and coma free days | while in ICU, appoximately 3-7 days)
Incidence of subacute cognitive dysfunction using RBANS- Repeatable Battery for the Assessment of Neuropsychological Status, | 3 months
Incidence of subacute cognitive dysfunction using TRAILS A&B | 3 months
Incidence of subacute cognitive dysfunction using SF-36 - Short Form Health Survey | 3 months
Incidence of subacute cognitive dysfunction using MMSE - Mini Mental State Examination | 3 months
Incidence of subacute cognitive dysfunction using IADLs - instrumental activities of daily living | 3 months
Incidence of subacute cognitive dysfunction using AD8- ADL - activities of daily living | 3 months
Incidence of subacute cognitive dysfunction using APACHE II - Acute Physiologic and Chronic Health Evaluation II score | 3 months
ICU length of stay | while in ICU, appoximately 3-7 days
Hospital length of stay | while in hospital, usually 5-10 days
Six month mortality | 6 months
Biomarkers for neurological injury and inflammation, Neuron-Specific Enolase (NSE) | Baseline, Day 3 and at Ventilator removal (appoximately day 3-7)
Biomarkers for neurological injury and inflammation, S100 | Baseline, Day 3 and at Ventilator removal (appoximately day 3-7)
Biomarkers for neurological injury and inflammation, IL-6 | Baseline, Day 3 and at Ventilator removal (appoximately day 3-7)
Biomarkers for neurological injury and inflammation, C Reactive Protein (CRP) | Baseline, Day 3 and at Ventilator removal (appoximately day 3-7)
sleep quality | within 24 hours of enrollment through day 3-7
  measured with continuous polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Wes Ely, MD, Principal Investigator — Vanderbilt Universtiy
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Marcantonio ER, Juarez G, Goldman L, Mangione CM, Ludwig LE, Lind L, Katz N, Cook EF, Orav EJ, Lee TH. The relationship of postoperative delirium with psychoactive medications. JAMA. 1994 Nov 16;272(19):1518-22. PMID 7966844
- [Background] Pandharipande P, Shintani A, Peterson J, Pun BT, Wilkinson GR, Dittus RS, Bernard GR, Ely EW. Lorazepam is an independent risk factor for transitioning to delirium in intensive care unit patients. Anesthesiology. 2006 Jan;104(1):21-6. doi: 10.1097/00000542-200601000-00005. PMID 16394685
- [Background] Inouye SK, Schlesinger MJ, Lydon TJ. Delirium: a symptom of how hospital care is failing older persons and a window to improve quality of hospital care. Am J Med. 1999 May;106(5):565-73. doi: 10.1016/s0002-9343(99)00070-4. PMID 10335730
- [Background] Dubois MJ, Bergeron N, Dumont M, Dial S, Skrobik Y. Delirium in an intensive care unit: a study of risk factors. Intensive Care Med. 2001 Aug;27(8):1297-304. doi: 10.1007/s001340101017. PMID 11511942
- [Background] Inouye SK, Charpentier PA. Precipitating factors for delirium in hospitalized elderly persons. Predictive model and interrelationship with baseline vulnerability. JAMA. 1996 Mar 20;275(11):852-7. PMID 8596223
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Milbrandt EB, Deppen S, Harrison PL, Shintani AK, Speroff T, Stiles RA, Truman B, Bernard GR, Dittus RS, Ely EW. Costs associated with delirium in mechanically ventilated patients. Crit Care Med. 2004 Apr;32(4):955-62. doi: 10.1097/01.ccm.0000119429.16055.92. PMID 15071384
- [Background] Jackson JC, Gordon SM, Hart RP, Hopkins RO, Ely EW. The association between delirium and cognitive decline: a review of the empirical literature. Neuropsychol Rev. 2004 Jun;14(2):87-98. doi: 10.1023/b:nerv.0000028080.39602.17. PMID 15264710
- [Background] Jacobi J, Fraser GL, Coursin DB, Riker RR, Fontaine D, Wittbrodt ET, Chalfin DB, Masica MF, Bjerke HS, Coplin WM, Crippen DW, Fuchs BD, Kelleher RM, Marik PE, Nasraway SA Jr, Murray MJ, Peruzzi WT, Lumb PD; Task Force of the American College of Critical Care Medicine (ACCM) of the Society of Critical Care Medicine (SCCM), American Society of Health-System Pharmacists (ASHP), American College of Chest Physicians. Clinical practice guidelines for the sustained use of sedatives and analgesics in the critically ill adult. Crit Care Med. 2002 Jan;30(1):119-41. doi: 10.1097/00003246-200201000-00020. No abstract available. PMID 11902253
- [Background] Kollef MH, Levy NT, Ahrens TS, Schaiff R, Prentice D, Sherman G. The use of continuous i.v. sedation is associated with prolongation of mechanical ventilation. Chest. 1998 Aug;114(2):541-8. doi: 10.1378/chest.114.2.541. PMID 9726743
- [Background] Kress JP, Pohlman AS, O'Connor MF, Hall JB. Daily interruption of sedative infusions in critically ill patients undergoing mechanical ventilation. N Engl J Med. 2000 May 18;342(20):1471-7. doi: 10.1056/NEJM200005183422002. PMID 10816184
- [Background] Aurell J, Elmqvist D. Sleep in the surgical intensive care unit: continuous polygraphic recording of sleep in nine patients receiving postoperative care. Br Med J (Clin Res Ed). 1985 Apr 6;290(6474):1029-32. doi: 10.1136/bmj.290.6474.1029. PMID 3921096
- [Background] Cooper AB, Thornley KS, Young GB, Slutsky AS, Stewart TE, Hanly PJ. Sleep in critically ill patients requiring mechanical ventilation. Chest. 2000 Mar;117(3):809-18. doi: 10.1378/chest.117.3.809. PMID 10713011
- [Background] Sleigh JW, Andrzejowski J, Steyn-Ross A, Steyn-Ross M. The bispectral index: a measure of depth of sleep? Anesth Analg. 1999 Mar;88(3):659-61. doi: 10.1097/00000539-199903000-00035. PMID 10072023
- [Background] Grocott HP, Newman MF, El-Moalem H, Bainbridge D, Butler A, Laskowitz DT. Apolipoprotein E genotype differentially influences the proinflammatory and anti-inflammatory response to cardiopulmonary bypass. J Thorac Cardiovasc Surg. 2001 Sep;122(3):622-3. doi: 10.1067/mtc.2001.115152. No abstract available. PMID 11547323
- [Background] Weigand MA, Volkmann M, Schmidt H, Martin E, Bohrer H, Bardenheuer HJ. Neuron-specific enolase as a marker of fatal outcome in patients with severe sepsis or septic shock. Anesthesiology. 2000 Mar;92(3):905-7. doi: 10.1097/00000542-200003000-00057. No abstract available. PMID 10719986
- [Background] Hopkins RO, Weaver LK, Pope D, Orme JF, Bigler ED, Larson-LOHR V. Neuropsychological sequelae and impaired health status in survivors of severe acute respiratory distress syndrome. Am J Respir Crit Care Med. 1999 Jul;160(1):50-6. doi: 10.1164/ajrccm.160.1.9708059. PMID 10390379
- [Background] Norris PR, Dawant BM. Closing the loop in ICU decision support: physiologic event detection, alerts, and documentation. Proc AMIA Symp. 2001:498-502. PMID 11825238
- See also: This is an educational website about ICU delirium. — http://www.ICUdelirium.org